CLINICAL TRIAL: NCT04303585
Title: Blocco Del Dentato Anteriore e Blocco Del Muscolo Erettore Della Colonna Vertebrale Nella Gestione Multimodale Del Dolore in Chirurgia Toracica Mininvasiva: Studio Osservazionale Prospettico Multicentrico
Brief Title: SAP Versus ESP Block in Multimodal Pain Management in Mini-invasive Thoracic Surgery: an Observational Prospective Multicentric Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Trieste (Other)
Collaborators: Cliniche Humanitas Gavazzeni (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other)
Responsible Party: Principal Investigator, Marzia Umari, Principal Investigator, University of Trieste
Other Study IDs: 145_2018 Blocco gran dentato
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: SAP Block Versus ESP Block; Pain, Postoperative; Evaluation of Locoregional Techniques; Multimodal Pain Management
Keywords: SAP block; ESP block; Pain management; Mini-invasive; Thoracic surgery; SAP; ESP; Locoregional; Multimodal
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SAP block: This group includes patients who receive preoperative Serratus Anterior Plane block
  Interventions: Procedure: SAP block
- ESP block: This group includes patients who receive preoperative Erector Spinae Plane block
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: SAP block — The anesthesiologist performs SAP block immediately before surgery under ultrasound guide
  Groups: SAP block
Procedure: ESP block — The anesthesiologist performs ESP block immediately before surgery under ultrasound guide
  Groups: ESP block

SUMMARY:
Thoracic surgery is characterized by acute perioperative pain. There are different ways to provide analgesia, such as intravenous analgesics (opioids or non-opioids) or loco-regional procedures; these techniques are often used together in the context of a multimodal approach to pain management, in order to exploit their synergistic action and minimize side effects. In this observational prospective multicentric study the investigators evaluate the effectiveness of two routinely administered ultrasound guided loco-regional analgesic techniques in providing analgesia to patients undergoing mini-invasive lung-resective thoracic surgery. The two techniques compared are the serratus anterior plane (SAP) block and the erector spinae plane (ESP) block.

DETAILED DESCRIPTION:
Whatever the loco-regional technique is (SAP block or ESP block), it must have been administered in the immediate preoperative phase; both procedures are routinely used for analgesic purpose in the clinical practice of the three centers involved in the study and are performed under ultrasound guide. Using medical records, data collected by Acute Pain Service nurses and patients' interviews useful data will be collected: demographic and clinical characteristics (age, sex, weight, comorbidities), surgical data (type of procedure, surgical approach and duration of surgery) and anesthesia data (type of block, dose and type of local anesthetic with record of potential side effects), intraoperative and postoperative opioid and non-opioid analgesic consumption (and rescue if needed) with record of potential side effects, pain evaluation in the first 24 hours after surgery and after at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Lung-resective thoracic surgery (lobectomy, bilobectomy, segmentectomy and wedge resection) with videothoracoscopic or mini-thoracotomic approach (maximum duration 180 minutes)
* BMI ranging from 18 to 30
* Age > 18 years
* ASA I-III
* Ultrasound guided preoperative ESP block or SAP block
* Remifentanil as intraoperative opioid

Exclusion Criteria:

* Patient's refusal
* Weight < 50 kg
* Pregnancy
* Emergent surgery
* Chronic opioid therapy
* History of drug or benzodiazepine addiction or alcohol abuse
* Previous thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized in one of the centers taking part in the study undergoing mini-invasive lung-resective thoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | First 24 hours after surgery
  Evaluation of morphine consumption in the first 24 hours after surgery

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Duration of surgical procedure
  Evaluation of opioid consumption during lung-resective thoracic surgery
Numeric Rating Scale (NRS) | First 24 hours after surgery, then after 3 months
  Evaluation of NRS for static, dynamic and cough-associated pain
Analgesic rescue and corticosteroids | First 24 hours after surgery
  Evaluation of eventual administration of rescue analgesic drugs and corticosteroids in the first 24 hours after surgery
Side effects | First 24 hours after surgery
  Evaluation of eventual side effects related to the locoregional techinque or the analgesics used (LAST, hypotension, Post Operative Nausea and Vomiting (PONV) and opioid-related side effects) in the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Lucangelo, MD PhD, Study Chair — University of Trieste; Marzia Umari, MD, Principal Investigator — University of Trieste; Giovanni Albano, MD, Principal Investigator — Cliniche Humanitas Gavazzeni; Edoardo Ceraolo, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza - Molinette Hospital
Locations (3):
- Italy (3):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - A.O.U. Città della Salute e della Scienza - Molinette Hospital, Torino
  - Cattinara Hospital, Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okmen K, Okmen BM. The efficacy of serratus anterior plane block in analgesia for thoracotomy: a retrospective study. J Anesth. 2017 Aug;31(4):579-585. doi: 10.1007/s00540-017-2364-9. Epub 2017 Apr 26. PMID 28447227
- [Background] McGovern I, Walker C, Cox F. Pain relief after thoracotomy. Br J Anaesth. 2007 Jun;98(6):844; author reply 844-5. doi: 10.1093/bja/aem112. No abstract available. PMID 17519266
- [Background] Wenk M, Schug SA. Perioperative pain management after thoracotomy. Curr Opin Anaesthesiol. 2011 Feb;24(1):8-12. doi: 10.1097/ACO.0b013e3283414175. PMID 21084984
- [Background] Doan LV, Augustus J, Androphy R, Schechter D, Gharibo C. Mitigating the impact of acute and chronic post-thoracotomy pain. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):1048-56. doi: 10.1053/j.jvca.2014.02.021. No abstract available. PMID 25107721
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192
- [Background] Luis-Navarro JC, Seda-Guzman M, Luis-Moreno C, Lopez-Romero JL. The erector spinae plane block in 4 cases of video-assisted thoracic surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Apr;65(4):204-208. doi: 10.1016/j.redar.2017.12.004. Epub 2018 Jan 11. English, Spanish. PMID 29336785
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Scimia P, Basso Ricci E, Droghetti A, Fusco P. The Ultrasound-Guided Continuous Erector Spinae Plane Block for Postoperative Analgesia in Video-Assisted Thoracoscopic Lobectomy. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):537. doi: 10.1097/AAP.0000000000000616. No abstract available. PMID 28632673
- [Background] Rao Kadam V, Currie J. Ultrasound-guided continuous erector spinae plane block for postoperative analgesia in video-assisted thoracotomy. Anaesth Intensive Care. 2018 Mar;46(2):243-245. No abstract available. PMID 29519230
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Leyva FM, Mendiola WE, Bonilla AJ, Cubillos J, Moreno DA, Chin KJ. Continuous Erector Spinae Plane (ESP) Block for Postoperative Analgesia after Minimally Invasive Mitral Valve Surgery. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2271-2274. doi: 10.1053/j.jvca.2017.12.020. Epub 2017 Dec 12. No abstract available. PMID 29336964
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621